# Outcomes of Metabolic Resuscitation Using Ascorbic Acid, Thiamine, and Glucocorticoids in the Early Treatment of Sepsis.

### **ORANGES Trial**

NCT#: NCT03422159

Document Date: May 13<sup>th</sup>, 2019

## Study end-points:

## **Primary end-point**

- i. Time to vasopressor independence. Defined as the time from starting the active treatment/placebo to discontinuation of all pressors
- ii. Delta SOFA score, defined as the initial SOFA score minus the day 4 SOFA score

### **Secondary end-points**

- iii. 28-day mortality
- iv. Hospital mortality
- v. PCT clearance (PCT-c) calculated using the following formula: initial PCT minus PCT at 96 hours, divided by the initial PCT multiplied by 100. [67,68]
- vi. ICU mortality
- vii. ICU length of stay (LOS) and ICU free days. ICU free days is calculated as the number of days alive and out of the ICU to day 28
- viii. Hospital LOS

## **Power Calculation:**

Based on the results of the preliminary study of Marik et al we project that the combination of hydrocortisone, vitamin C and thiamine could reduce time to vasopressor discontinuation from 54 (+/-30 hours) versus 30 hours. For the additional primary outcome we projected a greater change of SOFA

score of 4 (+/- 3) versus 2. Assuming a type 1 error of 5% (alpha of 0.05) and a power of 80% (the ability to detect a difference between two groups when a difference exists) would require a sample size of 94 patients. To account for dropouts and patients not requiring vasopressor therapy we will therefore aim for a sample size of 140 patients.

## Data analysis:

Summary statistics will be used to describe the clinical data and presented as mean  $\pm$  SD, median with interquartile range (IQR) or percentages as appropriate. Chi squared analysis with Fisher's exact test (when appropriate) and Student's t test (Mann Whiney U test for non- normal distributions) were used to compare data between the active treatment group and the placebo group with statistical significance declared for probability values of 0.05 or less.